CLINICAL TRIAL: NCT00426569
Title: Normal Paranasal Sinuses Microflora Study
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Arkadi Yakirevitch, Arkadi Yakirevitch, MD, Sheba Medical Center
Other Study IDs: SHEBA-07-4534-AY-CTIL
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Paranasal Sinuses; Flora

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to check if bacterial and fungal flora exists in healthy paranasal sinuses, and whether it is identical to the flora of nasal cavity.

We plan to harvest tiny examples of maxillary sinus and nasal mucosa for tissue cultures during the orthognathic procedures involving maxillary remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Necessity of maxillary sinus opening during orthognathic surgery
* Negative history of chronic rhinitis or chronic sinusitis
* Informed concent

Exclusion Criteria:

* Recent(1 month or less before the operation) event of acute sinusitis or other disease leading to nasal discharge
* Recent(1 month or less before the operation) antibacterial or antifungal parenteral treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy adults undergoing orthognatic procedure
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-02; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
presence of bacteria in normal paranasal sinuses | at time of orthgnatic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arkadi Yakirevitch, M.D., Principal Investigator — Department of Otorhinolaryngology-Head and Neck Surgery, Sheba Medical Center, Israel
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel